CLINICAL TRIAL: NCT04543604
Title: Understanding, Modulation and Memorization of Indicators Associated to Peri-implantitis: A Randomized Controlled Trial
Brief Title: Understanding, Modulation and Memorization of Indicators Associated to Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18002909-18/9/19
Record Dates: First submitted 2020-08-29; First posted 2020-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Audiovisual Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group1 - Leaflet with visual aid (Experimental): Information concerning etiology, prevalence, risk indicators and preventive measures of peri-implantitis were included. Relevant scientific bibliography supported the statements. Along, pictograms were supplemented to display the prevalence of disease with and without the known indicator.
  Interventions: Behavioral: Leatlet + visual aid (pictogram)
- Test group2 - Leaflet with visual aid (L-NVA) (Experimental): Information concerning etiology, prevalence, risk indicators and preventive measures of peri-implantitis were included. Relevant scientific bibliography supported the statements. No pictograms were supplemented.
  Interventions: Behavioral: Leaflet + no visual aid (no pictogram)
- • Control group - No leaflet (NL) (No Intervention): Only verbal information was provided to the patient during initial interview.

INTERVENTIONS:
Behavioral: Leatlet + visual aid (pictogram) — The questionnaires were collected at baseline (at the end of the initial interview and once the patients assigned within the test groups declared to have read the leaflet) at 3- and 6-month follow-up. The questionnaire included demographic data such as age, gender, civil status, occupation (coded according to the CNO-11(2010), presence of systemic disorder, smoking and number of implants. Moreover, data concerning history of periodontal disease and type of prosthesis were further documented and added to demographics.
  Arms: Test group1 - Leaflet with visual aid
Behavioral: Leaflet + no visual aid (no pictogram) — The questionnaires were collected at baseline (at the end of the initial interview and once the patients assigned within the test groups declared to have read the leaflet) at 3- and 6-month follow-up. The questionnaire included demographic data such as age, gender, civil status, occupation (coded according to the CNO-11(2010), presence of systemic disorder, smoking and number of implants. Moreover, data concerning history of periodontal disease and type of prosthesis were further documented and added to demographics.
  Arms: Test group2 - Leaflet with visual aid (L-NVA)

SUMMARY:
Communication strategies are encouraged to enhance patients´ understanding of potential events related to implant therapy such as peri-implantitis. Moreover, it is key to provide accurate information to patients receiving dental implants to reduce false expectations and to minimize the alterations concerning satisfaction. Information leaflets based in the "health-belief model" proved efficiency in improving health judgments, decisions and behaviors, in particular when supplemented with visual aids. Hence, it was the purpose of the present study to test the effectiveness of different communication strategies to enhance and modulate the understanding and memorization of risk indicators associated to peri-implantitis.

A prospective randomized controlled three-arm study is being conducted in accordance with the Declaration of Helsinki on human studies. Three groups are defined to test the hypothesis that visual aids improve the understanding, modulation and memorization of peri-implantitis and related indicators as follows:

* Test group1 - Leaflet with visual aid (L-VA): Information concerning etiology, prevalence, risk indicators and preventive measures of peri-implantitis were included (supplementary figure 1). Relevant scientific bibliography supported the statements. Along, pictograms were supplemented to display the prevalence of disease with and without the known indicator.
* Test group2 - Leaflet with visual aid (L-NVA): Information concerning etiology, prevalence, risk indicators and preventive measures of peri-implantitis were included (supplementary figure 2). Relevant scientific bibliography supported the statements. No pictograms were supplemented.
* Control group - No leaflet (NL): Only verbal information was provided to the patient during initial interview.

Patients will be randomly assigned to the tests or control groups according to the last digit of their chart number. As such, patients with records ending 1-4, 4-7 and 8-0 were included in test group1, test group2 and control group, respectively. When reached the total sample size of any of the groups, patients were only recruited for the remaining groups to complete the total sample size. A questionnaire based on the "health-belief model" will be collected from every eligible patient at baseline, 3- and 6-month follow-up

ELIGIBILITY:
The following inclusion criteria were applied: partially or completely edentulous patients aged 18-80 years and rehabilitated with implant-supported, single-crown fixed prostheses or implant-supported overdentures; smokers or non-smokers; absence of infectious disease at the time of implant placement; and absence of systemic disorders or medications known to alter bone metabolism. Subjects were excluded if they were pregnant; presented uncontrolled medical conditions or diseases (i.e., diabetes mellitus with HbA1c level >8); or presented zygomatic or pterygoid implants. Patients with treated peri-implantitis/mucositis were likewise excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Understanding | Baseline
  Questionnaire
Memorisation | 3 month follow-up
  Questionnaire
Memorisation | 6 month follow-up
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Implantologia Cirugia Oral y Maxilofacial, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Monje A, Perez A, Vera-Rodriguez M, Nart J, Catena A, Petrova D. Comprehension and recall of information about factors associated with peri-implantitis: A randomized controlled trial. J Periodontol. 2022 Jan;93(1):89-99. doi: 10.1002/JPER.21-0018. Epub 2021 May 27. PMID 33949680